CLINICAL TRIAL: NCT04455295
Title: Testing the Noradrenergic Hypothesis of Transcutaneous Vagus Nerve Stimulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Roosevelt_102218
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: no Condition; Electroencephalography; Pupil Diameter

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Stimulation 0.5 (Experimental): 0.5mA, 30Hz intermittent transdermal vagus nerve stimulation of the auricle vagus. Stimulation 30 second on/30 seconds off for five cycles.
  Interventions: Device: Transdermal Vagus Nerve Stimulation (tVNS)
- Lobe Control (Placebo Comparator): 0.5mA, 30Hz intermittent transdermal vagus nerve stimulation of the earlobe. Stimulation 30 second on/30 seconds off for five cycles.
  Interventions: Device: Transdermal Vagus Nerve Stimulation (tVNS)
- Sham Stimulation (Placebo Comparator): 0.5mA, 5Hz intermittent transdermal vagus nerve stimulation of the auricle vagus. Stimulation 30 second on/30 seconds off for five cycles.
  Interventions: Device: Transdermal Vagus Nerve Stimulation (tVNS)
- Nonstimulation (Placebo Comparator): Placement of electrode without any stimulation.
  Interventions: Device: Transdermal Vagus Nerve Stimulation (tVNS)

INTERVENTIONS:
Device: Transdermal Vagus Nerve Stimulation (tVNS) — Mild non-invasive transdermal electrical stimulation at the ear (0.0-1.0 mA, 0.0-30.0 Hz). Used in previous studies with no unexpected adverse events. Stimulator not considered a FDA regulated device in previous studies.

SUMMARY:
This study investigates the capacity of non-invasive vagus nerve stimulation, applied at the ear, to alter to measures of locus coeruleus output pupil diameter and EEG alpha power. Non-invasive alteration in locus coeruleus output is of interest in regard to basic science and has potential clinical implications in a number of conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, 18 years of age or older.

Exclusion Criteria:

* self-report of mood disorders, prescription and non-prescription drug use which includes stimulants including caffeine and nicotine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Pupil Diameter | Within single one hour session
  Pupil diameter is measured via camera.
EEG Alpha power. | Within single one hour session
  Alpha power will be determined from EEG.

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Tech University, Russellville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT04455295/Prot_SAP_ICF_000.pdf